CLINICAL TRIAL: NCT03312114
Title: Phase II Trial of Concurrent Anti-PD-L1 and SAbR for Patients With Persistent or Recurrent Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancer (With Safety lead-in)
Brief Title: Anti-PD-L1 and SAbR for Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 032017-078
Record Dates: First submitted 2017-09-14; First posted 2017-10-17 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Recurrent Epithelial Cancer of Ovary; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Avelumab and SABR
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab* (MSB0010718C; anti-PD-L1 is a fully human anti-PD- L1 IgG1 antibody)
  Other Names: Bavencio

SUMMARY:
Programmed death-1 receptor ligand (PD-L1) the ligand for PD-1 is a key therapeutic target in the reactivation of the immune response against multiple cancers. Pharmacologic inhibitors of PD-1 have also demonstrated significant anti-tumor activity and are currently under active clinical exploration. avelumab (MSB0010718C; anti-PD-L1 is a fully human anti-PD-L1 igG1 antibody that has shown promising efficacy and an acceptable safety profile in multiple tumor types.

Radiation therapy (RT) is one of the mainstream treatments of cancer therapy along with surgery and chemotherapy, yet RT is the only treatment that does not leave the patients immunocompromised (unlike chemotherapy) and keeps the dying tumor / antigen depot within the host (unlike surgery), providing an opportunity for antigen presentation. Therefore, RT is a rational choice to combine with immunotherapy for cancer treatment.

DETAILED DESCRIPTION:
Screening/Baseline Procedures Assessments performed exclusively to determine eligibility for this study will be done only after obtaining informed consent. Assessments performed for clinical indications (not exclusively to determine study eligibility) may be used for baseline values even if the studies were done before informed consent was obtained.

All screening procedures must be performed within 28 days prior to registration unless otherwise stated. The screening procedures include:

* Informed Consent
* Medical history: Complete medical and surgical history, history of infections
* Demographics: Age, gender, race, ethnicity
* Review subject eligibility criteria
* Review previous and concomitant medications
* Physical exam including vital signs, height and weight: Vital signs (temperature, pulse, respirations, blood pressure), height, weight
* Performance status: Performance status evaluated prior to study entry according to Appendix #/letter.
* Adverse event assessment: Baseline adverse events will be assessed. See section 6 for Adverse Event monitoring and reporting.
* Hematology CBC and diff ( within 2 weeks of registration)
* T 4 levels, TSH and CMP as below: Comprehensive metabolic panel (CMP) to include: albumin, alkaline phosphatase, ALT/SGPT, AST/SGOT, BUN, creatinine, electrolytes (sodium, potassium, calcium, chloride, bicarbonate), glucose, and total bilirubin. (within 2 weeks of registration)- Pregnancy test (for females of child bearing potential)( within 2 weeks of registration)
* Tumor assessment:Baseline imaging by CT scan of chest , abdomen, and pelvis.

Procedures During Treatment

* Prior to Each Treatment Cycle

  * Physical exam, vital signs
  * Hematology
  * Serum chemistries
* Every 8 weeks after start till end of treatment Serum TSH, pregnancy test and CT chest abdomen and pelvis

  30 days after treatment termination
* Physical exam, vital signs
* Hematology
* Serum chemistries
* additional Immune co-relate lab testing: Prior to cycle 1, cycle 3, cycle 5, cycle 7 and 2 weeks post last cycle.

Follow-up Procedures

* For patients who are still receiving Avelumab: Subject will be followed every eight weeks (+/- 2 weeks) starting from the beginning of treatment for the first year, then every 12 weeks (+/- 2 weeks) till 2 years after last dose of drug The following procedures will be performed at each follow up:

  * Physical exam, PS, vital signs, medication review, AE assessment
  * Blood collection per time table and for labs
  * Radiographic imaging: Tumor assessments will be completed by the investigator using the RECIST criteria as above.

    * CT chest, abdomen and pelvis with IV contrast, if allowable by renal function
    * After that, survival information will be collected every 6 months until patient death.
* For patients who have been discontinued from Avelumab : Subject will be followed 30 days from last dose (±7 days, or may be on date of discontinuation ±7 days if the date of discontinuation is more than 37 days after last dose) and then 3-4 months from last dose.

The following procedures will be performed at the first two visits:

* Physical exam, PS, vital signs, medication review, AE assessment
* Subsequent anti-cancer treatment/s
* For first visit only, or may repeat if study drug related toxicity persists: CBC w/ differential, LFTs, BUN, creatinine, fasting glucose, and TSH

After that, survival information will be collected every 6 months until patient death.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged ≥ 18 years.
2. Performance ECOG status of 0-2
3. Patient is able and willing to comply with protocol and study procedures for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up visits.
4. Adequate Physiologic function:

   * Hematologic: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused)
   * Hepatic: Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
   * Renal: Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
5. Pregnancy and contraception:

   Pregnancy test: Negative serum or urine pregnancy test at screening for women of childbearing potential.

   Contraception: Women of child-bearing potential and their male partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry.,
6. Histologic diagnosis of recurrent epithelial ovarian ,fallopian ,peritoneal cancer
7. Patients with platinum sensitive ovarian cancer must have progressed through at least one platinum containing regimen for recurrent disease.
8. Patients with platinum resistant ovarian cancer must have progressed through at least one prior chemotherapy regimen for recurrent ovarian cancer.
9. Patients must have received at least one prior chemotherapy regimen and up to any number of prior systemic regimens including chemotherapy and molecular targeted therapy other than PD1/ PDL1/ PDL2 inhibitors.
10. Metastatic disease of at least two Non-CNS sites (including the index lesion to be treated) measurable by RECIST criteria with at least one site outside of the radiation field and evaluable by RECIST criteria for evaluation of response.
11. Ability to understand and the willingness to sign a written informed consent -

Exclusion Criteria:

1. IMMUNOSUPRESSANTS: "Current use of immunosuppressive medication, EXCEPT for the following: a. Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)."
2. AUTOIMMUNE DISEASE: "Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible."
3. ORGAN TRANSPLANTATION: "Prior organ transplantation including allogenic stem-cell transplantation."
4. HIV/AIDS: "Known history of testing positive for HIV or known acquired immunodeficiency syndrome."
5. HEPATITIS: "Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)"
6. VACCINATION: "Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines "
7. HYPERSENSITIIVTY TO STUDY DRUG: "Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)"
8. CARDIOVASCULAR DISEASE: "Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication."
9. OTHER PERSISTING TOXICITIES: "Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 2); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable."
10. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis ,Severe COPD requiring > 3 hospitalization in the past year Or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
11. No concomitant therapy with any of the following: IL2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; or other investigational therapies; all such therapies must have been discontinued >4weeks prior to registration.
12. No active TB,
13. Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy.
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Patients must not be pregnant or nursing.
16. No history of prior treatment with inhibitor of PD-1 or PD-L1 or PDL2.
17. Major surgery within 2 weeks prior to registration or first dose of drug
18. Subjects who have had radiation therapy within 2 weeks prior to first dose of drug
19. Uncontrolled adrenal insufficiency or active chronic liver disease
20. Any history of CNS metastases that is not adequately treated (surgery or radiation ) >14 days prior to registration.
21. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalent are permitted (although not encouraged) in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects aged ≥ 18 years.
Enrollment: 5 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Albuquerque, MD, Principal Investigator — kevin.albuquerque@utsouthwestern.edu
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Avelumab and SABR
  Trial of combined Avelumab with SAbR for Recurrent Ovarian and peritoneal, fallopian tube cancer (ROPT) is to assess overall clinical response rates per RECIST criteria.
Period: Overall Study
Arm/Group | Single Arm
Started | 5
Completed | 0
Not Completed | 5
Not completed — All the five enrolled dropped out of the | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 63 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: data was not analyzed
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: To Assess Overall Clinical Response Rates Per RECIST Criteria.
Description: Analysis of (with safety lead-in) trial of combined Avelumab (MSB0010718C) anti-PD-L1checkpoint blockade with SAbR for Recurrent Ovarian and peritoneal ,fallopian tube cancer (ROPT) is to assess overall clinical response rates per RECIST criteria .
Time Frame: 1 year,4 months
Population: All patients progressed- without any response.
Measure: Count of Participants; unit: Participants
Groups:
- Recurrent Ovarian and Peritoneal ,Fallopian Tube Cancer (ROP: The primary objective of this phase II(with safety lead-in) trial of combined Avelumab (MSB0010718C) anti-PD-L1checkpoint blockade with SAbR for Recurrent Ovarian and peritoneal ,fallopian tube cancer (ROPT) is to assess overall clinical response rates per RECIST criteria . This will be after the safety lead-in is completed without DLT at 8 weeks from start of Avelumab, to evaluate the safety of Avelumab and SABR to an acceptable dose of the site radiated.
Arm/Group | Recurrent Ovarian and Peritoneal ,Fallopian Tube Cancer (ROP
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Overall Survival
Description: Patients were started on alternative therapy and were not followed after starting alternative therapy.
  Study was stopped because drug was found to be ineffective by the pharmaceutical company
Time Frame: 1 year, 4 months
Population: All the five enrolled dropped out of the study early due to disease progression.
  Study was stopped because drug was found to be ineffective by the pharmaceutical company.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 5
Participants | NA — All the five enrolled dropped out of the study early due to disease progression. Study was stopped because drug was found to be ineffective by the pharmaceutical company

ADVERSE EVENTS:
Time Frame: The adverse event were 6 months from enrollment
Groups:
- Concurrent Anti-PD-L1 + SAbR to Metastasis: There were no serious adverse events on the trial.
Arm/Group | Concurrent Anti-PD-L1 + SAbR to Metastasis
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Anti-PD-L1 + SAbR to Metastasis (N=5)
LYMPHOCYTE COUNT DECREASED (Blood and lymphatic system disorders) | 5 (7)
FATIGUE (General disorders) | 5 (6)
CONSTIPATION (Gastrointestinal disorders) | 5 (6)
ANOERXIA (General disorders) | 5 (5)
VOMITING (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT03312114/Prot_SAP_000.pdf